CLINICAL TRIAL: NCT00988936
Title: A Phase II, Open Label, Non-randomized, Multi-center, Pilot, Efficacy Study of [F-18]RGD-K5 Positron Emission Tomography (PET) as a Tool to Monitor Response to an Anti-angiogenic Drug
Brief Title: Efficacy Study of [F-18]RGD-K5 Positron Emission Tomography (PET) as a Tool to Monitor Response to an Anti-angiogenic Drug
Acronym: K5-101
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Siemens Molecular Imaging (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: K5-101
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Metastatic Breast Cancer; Metastatic Colon/Rectum Cancer; Non-squamous Non-small Cell Lung Cancer
Keywords: [F-18]RGD-K5; RGD-K5; K5-101; Avastin; angiogenesis; anti-angiogenesis; chemotherapy; breast cancer; colon cancer; rectal cancer; lung cancer; non-squamous; non small cell
MeSH Terms: conditions — Breast Neoplasms; Rectal Neoplasms; Colonic Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [F-18]RDG-K5 (Experimental)
  Interventions: Drug: [F-18]RGD-K5

INTERVENTIONS:
Drug: [F-18]RGD-K5 — Approximately forty (40) patients with non-squamous non-small cell lung cancer, metastatic breast cancer, metastatic colon or rectum cancer will receive chemotherapy plus Avastin® and will be imaged under PET/CT with [F-18]RGD-K5

SUMMARY:
A Pilot Phase II Study

The primary objective for this study is:

* To explore the usefulness of [F-18]RGD-K5 PET/CT to predict efficacy or early response to Avastin® (the anti-angiogenesis drug) plus chemotherapy treatment before the full course of treatment is completed

The secondary objectives for this study are:

* To continue safety evaluation by collection of safety data from all patients
* To gain experience with [F-18]RGD-K5 PET/CT in order to improve the study design and conduct of future studies

Design: An open label, non-randomized, uncontrolled, single group assignment, pilot efficacy study

Duration: Screening visit (3-4 hrs), pre-treatment imaging visit of [F-18]RGD-K5 PET/CT (~ 3-4 hrs) and the standard [F-18]FDG PET/CT (~ 3-4 hrs) or diagnostic CT, followed by two [F-18]RGD-K5 PET/CT scans, one after the second but before the third Avastin® treatment, and one after the fourth but before the fifth Avastin® treatment, and a follow up standard [F-18]FDG PET (~ 3-4 hrs) or diagnostic CT.

Procedures: Informed consent, collection of demographic information, medical history, blood labs, physical examination, vital signs, ECGs, three sets of [F-18]RGD-K5 dosing and imaging scans including pretreatment, early mid-treatment, and later mid-treatment, concomitant medication collection, adverse event monitoring, and assessment of tumor response to treatment

Patients: Approximately forty (40) patients with non-squamous non-small cell lung cancer, metastatic breast cancer, metastatic colon or rectum cancer who will receive chemotherapy plus Avastin®. This allows for approximately 30 evaluable patients to complete this study at approximately four to eight sites internationally

DETAILED DESCRIPTION:
The aim of this pilot study is to examine the utility of a new molecular imaging tracer, [F-18]RGD-K5 to monitor treatment responses in patients scheduled to undergo treatment with Avastin® (Bevacizumab) plus standard chemotherapy. The changes of [F-18]RGD-K5 PET/CT image scans between before treatment and after both mid-treatment cycles of Avastin® (Bevacizumab) will be evaluated. The hypothesis for this study is that changes in the uptake of [F-18]RGD-K5 PET in tumors may reflect changes in the level of integrin expression and/or angiogenesis. This pilot study will help to define if changes in uptake of [F-18]RGD-K5 are an early indicator of treatment efficacy to Avastin®.

ELIGIBILITY:
Inclusion Criteria:

* Patient is >18 years and male or female of any race / ethnicity
* Patient or patient's legally acceptable representative provides written informed consent and willing to comply with protocol requirements
* Patient must be scheduled to receive chemotherapy treatment(s) plus Avastin® for their cancer care; treatment management will be made by the treating medical oncologists (According to the package insert for Avastin®, it is administered as an IV infusion every 3 weeks for nonsquamous non-small cell lung cancer, and every 2 weeks for metastatic breast cancer, colon or rectum cancer)
* Patient will be scheduled to have a clinical [F-18]FDG-PET/CT or diagnostic CT pre-treatment after the fourth but before the fifth Avastin® treatment

Exclusion Criteria:

* Patient is not capable of complying with study procedures
* Female patient is pregnant or nursing; exclude the possibility of pregnancy by one of the following:

  * Confirming in medical history that the patient is postmenopausal for a minimum of one year, or surgically sterile
  * Confirming the patient is using one of the following methods of birth control for a minimum of one month prior to entry into this study: IUD, oral contraceptives, Depo-Provera, or Norplant
  * Confirming a negative urine dipstick test taken the morning of receiving the [F-18]RGD-K5
* Patient has a severe hepatic or renal disease as defined by previous medical history or abnormal renal and hepatic functions determined by lab results not within the following ranges, or in the opinion of the Investigator, the values are not acceptable for the patient to be included:

  * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limits of normal
  * Serum creatinine ≤ 2x institutional upper limits of normal
  * BUN within 2x institutional upper limits of normal
  * Patient has known hyper or hypo-coagulation syndromes. (e.g. Protein C, S deficiency, Hemophilia A/B/C, Factor-V Leiden, etc) or lab results are not within the following ranges, or in the opinion of the Investigator, the values are not acceptable for the patient to be included: Platelet counts of < 75 x 103/μL
* Patient has known sensitivity to any components of Avastin® such as recombinant human or humanized antibodies
* Patient has been involved in an investigative, radioactive research procedure within 7 days and during the study participation period
* Patient will participate in experimental therapy procedures while participating in this clinical trial
* Patient has any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete data or data quality to achieve study objectives, or complete study and/or post-dose follow-up examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-09; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To explore the usefulness of [F-18]RGD-K5 PET/CT to predict efficacy or early response to Avastin® (the anti-angiogenesis drug) plus chemotherapy treatment before the full course of treatment is completed. | (5) visits over a period of approximately 5 cycles of Avastin

SECONDARY OUTCOMES:
To continue safety evaluation by collection of safety data from all patients. | (5) visits over a period of approximately 5 cycles of Avastin
To gain experience with [F-18]RGD-K5 PET/CT in order to improve the study design and conduct of future studies. | (5) visits over a period of approximately 5 cycles of Avastin

CONTACTS AND LOCATIONS:
Overall Officials: Edward Aten, MD, Study Director — President, Certus International
Locations (8):
- United States (8):
  - University of California, Irvine, Irvine, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UMDNJ, Newark, New Jersey
  - Beth Israel Medical Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Hospital of University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Eastern Regional Medical Center, Philadelphia, Pennsylvania